CLINICAL TRIAL: NCT05822739
Title: A Single-Arm, Open-Label, Exploratory Clinical Study of BBM-P002 Gene Therapy for Parkinson's Disease
Brief Title: Safety and Efficacy Study of Parkinson's Disease Gene Therapy Drug (BBM-P002)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBM003- IIT1003
Record Dates: First submitted 2023-03-01; First posted 2023-04-21 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Gene therapy; Adeno-Associated Virus
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm of BBM-P002 (Experimental): single-arm
  Interventions: Drug: BBM-P002

INTERVENTIONS:
Drug: BBM-P002 — Genetic: single- dose intracranial injection of BBM-P002 Neurosurgical delivery of BBM-P002 to the brain
  Other Names: BBM003

SUMMARY:
Safety and Efficacy Study of BBM-P002 in participants with primary advanced Parkinson's disease

DETAILED DESCRIPTION:
Parkinson's disease is a neurodegenerative disorder involving loss of dopaminergic neurons in the substantia nigra. This study is a single-center, single-arm, open-label, treatment clinical study to evaluate the safety, tolerability and efficacy of an adeno-associated virus (AAV)-based gene therapy, termed BBM-P002, will be injected into the brain via a neurosurgical procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically confirmed diagnosis of idiopathic Parkinson's Disease (PD) in accordance with the 2015 Movement Disorder Society (MDS) diagnostic criteria.
2. Participants aged between 40 and 65 years, inclusive, of any gender.
3. A disease history of five years or more.
4. A Hoehn and Yahr (H-Y) stage of 2.5 to 4 in the Of-state.
5. An adeno-associated virus (AAV) neutralizing antibody titer of fit thecriteria.
6. A Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III score greater than 35 in the Off-state, with an improvement of at least 30% following an acute levodopa challenge test.
7. Stable anti-Parkinsonian medication regimen prior to the screening period for at least four weeks.
8. The subject must agree to postpone any other neurosurgical procedures (including deep brain stimulation) during the main study phase, with the exception of emergency neurosurgery for life-threatening conditions.
9. The subject must agree not to participate in other therapeutic interventional studies during the main study phase.
10. The subject must agree not to undergo vaccination during the main study phase.
11. Commitment to using a reliable method of contraception from the screening period until at least 52 weeks post-infusion.
12. The subject must be compliant and capable of attending regular follow-up appointments. The subject must be able to accurately complete a PD patient diary during the follow-up period, with assistance from family members, guardians, or caregivers permitted.
13. The subject must be fully informed about the nature, objectives, procedures, and potential adverse effects of the clinical trial, and must voluntarily consent to participate by signing the informed consent form. In cases where the subject is unable to read, a legally authorized representative or an impartial witness may read the informed consent form and other written materials to them and witness the consent process.

Exclusion Criteria:

1. Diagnosis of atypical or secondary parkinsonian syndromes (e.g., Parkinson-plus syndromes, hereditary parkinsonian syndromes, drug-induced parkinsonism).
2. Presence of surgical contraindications, a history of prior brain surgery such as deep brain stimulation (DBS), pallidotomy, or extrapyramidal surgery, or any other neurosurgical procedure that the investigator deems would interfere with participation in this trial.
3. Previous cranial imaging showing structural brain abnormalities, cerebrovascular malformations, intracranial tumors, risk of intracranial hemorrhage, traumatic brain injury, or other significant anomalies.
4. A Mini-Mental State Examination (MMSE) score of <24.
5. A Patient Health Questionnaire-9 (PHQ-9) score of ≥16.
6. Abnormal liver or kidney function, defined as: Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) >1.5 times the upper limit of normal (ULN), or serum creatinine (Cr) >1.5 times the ULN.
7. Coagulation dysfunction or current use of anticoagulant agents.
8. Positive screening for infectious diseases: positive for Hepatitis B surface antigen (HBsAg) or Hepatitis B virus DNA (HBV-DNA), positive for Hepatitis C virus RNA (HCV-RNA), positive for Human Immunodeficiency Virus (HIV), or seropositive for syphilis.
9. Currently undergoing antiviral treatment for Hepatitis B or C.
10. Presence of unstable or severe concomitant systemic diseases, including but not limited to active tuberculosis, or diseases of the cardiovascular, respiratory, digestive, urinary, neuropsychiatric (e.g., epilepsy), hematologic, or immune systems, or abnormal laboratory values that, in the judgment of the investigator, would make the subject unsuitable for the trial.
11. Current or prior history of a malignant tumor.
12. History of a severe allergic reaction, allergy to contrast agents, or inability to tolerate surgical anesthesia.
13. Current participation in another clinical trial, or participation in any other clinical trial within 3 months prior to the screening period.
14. Prior history of gene therapy before screening.
15. Receipt of stem cell therapy within 6 months prior to the screening period.
16. Use of other investigational drugs within 4 weeks prior to screening or within 5 half-lives of the drug (whichever is longer), or any medication judged by the investigator to interfere with the trial.
17. Receipt of a live vaccine within 2 months prior to the screening period, or any vaccination within 30 days prior to the screening period.
18. History of alcohol dependence or drug addiction, with an inability to adhere to medical advice to abstain from alcohol during the trial period.
19. Female subjectsparticipants who are pregnant or lactating.
20. Any subject deemed unsuitable for enrollment based on the investigator's assessment.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-04-14 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events and Serious Adverse Events | Day 1 through week 52
  Safety and Tolerability of BBM-P002 assessed by Adverse Events and Serious Adverse Event

SECONDARY OUTCOMES:
Efficacy of BBM-P002 | Change from Baseline to week 4，week 52
  Changes in gene expression product activity levels assessed by brain ¹⁸F-FDOPA PET
Efficacy of BBM-P002 | Change from Baseline to Week 52
  Changes in daily oral Levodopa (L-DOPA) dose or Levodopa Equivalent Dose (LEDD);
Efficacy of BBM-P002 | Change from Baseline to Week 52
  Changes in motor/no motor MDS-Unified Parkinson's Disease Rating Scale-Part III （UPDRS III) The UPDRS III score assesses motor symptoms of Parkinson's disease. The total score ranges from 0 to 132 points, with each of the 33 scoring points rated on a 5-point scale from 0 to 4. A score of 0 indicates normal, with no abnormalities. A score of 1 indicates mild, where symptoms are present but usually do not affect function. A score of 2 indicates mild, where symptoms are mild and have a minor impact on function. A score of 3 indicates moderate, where symptoms are moderate and have a significant impact on function. A score of 4 indicates severe, where symptoms are severe and lead to loss of function. The higher the score, the more severe the motor symptoms.
Efficacy of BBM-P002 | Change from Baseline to Week 52
  sleep disturbances were characterized using the Parkinson's Disease Sleep Scale-2 (PDSS-2) The PASS scale is a self-rating scale widely used internationally and specifically designed for patients with Parkinson's disease. It is used to systematically assess the occurrence frequency and severity of various sleep disorders in patients. There are a total of 15 items, each with a score range of 0 to 4 points, and a 5-level scoring method is adopted: 0 points: very mild/never (symptoms never occur or are very mild and do not cause disturbance) 1 point: Mild (symptoms occur occasionally and cause slight disturbance) · 2 points Moderate (symptoms occur frequently, moderate distress) · 3 points: Severe (symptoms occur frequently, severe distress) · 4 points: very severe/always (symptoms occur all the time or extremely severe). The score range is from 0 to 60 points. The higher the score, the more severe the sleep disorder.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai

IPD SHARING:
Plan to Share IPD: No